CLINICAL TRIAL: NCT07164599
Title: The Effects of 12-week Strength and Power Training on Movement Pattern, Physical Fitness and Lower Limb Strength Among Chinese College Sports Dancers
Brief Title: The Effects of 12-week Additional Strength Training and 8-week Detraining on Movement Patterns, Lower Limb Strength, and Dance Performance in Chinese College Dancesport Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Shazlin Shaharudin, Associate Professor, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: USM/JEPeM/KK/23040282
Record Dates: First submitted 2025-08-24; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers
Keywords: strength training; dancer; dancesport; muscle strength
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): strength training and dance traininig
  Interventions: Behavioral: strength training
- control group (No Intervention): dance training

INTERVENTIONS:
Behavioral: strength training — A 12-week strength training program designed for college dancesport athletes. Training is performed three times per week, 60 minutes per session, in addition to participants' regular dancesport training. Exercises include multi-joint resistance movements (e.g., squats, lunges, deadlifts, jumps) following NSCA guidelines with progressive overload based on 1RM. After the 12-week intervention, participants continue with an 8-week detraining phase without supplemental strength sessions and dance training.
  Arms: intervention group

SUMMARY:
In this study, which will investigate the effects of 12-week strength training with 8-week detraining on movement patterns, lower limb strength, and dance performance among Chinese college dancesport athletes, functional movement patterns, muscle architecture, lower limb strength and power, and dance performance will be measured. In dance activity, implementing appropriate strength conditioning programs can effectively enhance dancers' strength levels and improve performance while preserving the integrity of technical and aesthetic elements. The study is a randomized controlled trial. Dancesport major students will be assessed according to the screening conditions, and 30 participants will be recruited. Participants will be randomly assigned to an intervention group or a control group. The intervention group will undergo training three times per week, 60 minutes per session, for 12 weeks. All participants will undergo measurements at four time points: baseline, after six weeks, after twelve weeks, and after eight weeks of detraining.

DETAILED DESCRIPTION:
All participants are randomly allocated into the intervention group (n = 15) and the control group (n = 15). Allocation is performed by drawing lots. Fitness coaches and medical staff from Hubei Normal University who provide the intervention cannot be blinded to group allocation. The assessment staff remain unaware of the main group allocation. Participants are instructed to refrain from discussing their randomization assignment with the assessment staff or classmates. The study measurements include the functional movement screen, Y-balance test, lower limb muscle architecture, lower limb strength and power, and dance performance tests at baseline, mid-intervention, post-intervention, and after 8 weeks of detraining. During the intervention, training sessions are monitored using the rating of perceived exertion (RPE) and heart rate. Each complete measurement requires approximately two days. Written informed consent is obtained from all participants before the pre-intervention assessment. Day 1: muscle architecture, jump tests using a force platform, and dance performance test; Day 2: isokinetic strength tests, functional movement screen and Y-balance test. Before the first week of intervention, the research team demonstrates and teaches the participants the correct movement techniques, warm-up and stretching procedures, and baseline measurement procedures. Measurements are repeated after 6 and 12 weeks of intervention and after 8 weeks of detraining. The intervention group performs lower limb strength training for 12 weeks, three times per week, 60 minutes per session, in addition to dance training. The control group continues with dance training only, without any additional intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy women aged 18 years or older
2. Body mass index (BMI) between 18 and 28 according to the 2023 version of China's Physical Health Standard
3. At least 12 months of experience in dancesport training and learning
4. Participation in dancesport competitions at or above the city level
5. Voluntary agreement to participate in the study with provision of written informed consent

Exclusion Criteria:

1. Previous injuries that have not been rehabilitated, musculoskeletal injuries, or chronic pain
2. Exercise-related disorders, including coronary heart disease, peripheral vascular diseases, rhabdomyolysis, respiratory inflammation, neurological disorders, implanted electrical devices, or significant cognitive impairments
3. Current use of any medication or substance known to affect cardiorespiratory or metabolic responses to exercise, as described in Peel and Mossberg (1995)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-03-07 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Functional Movement Screen (FMS) Total Score | Baseline, 6 weeks, 12 weeks, and 8 weeks after detraining (up to 20 weeks per participant)
  Assesses fundamental movement quality using a standardized 7-action screening tool. The Functional Movement Screen (FMS) is a comprehensive tool designed to evaluate an individual's fundamental movement patterns. The FMS has been shown to correlate significantly with athletic performance, supporting its validity as a functional assessment tool.
Y-Balance Test | Baseline, 6 weeks, 12 weeks, and 8 weeks after detraining (up to 20 weeks per participant)
  The Y Balance Test is a validated functional assessment tool designed to evaluate dynamic balance, neuromuscular control, and injury risk in both upper and lower extremities by quantifying dynamic stability and identifying functional asymmetries predictive of lower extremity injury risk.
Isokinetic strength test for the knee and hip | Baseline, 6 weeks, 12 weeks, and 8 weeks after detraining (up to 20 weeks per participant)
  Isokinetic strength testing provides a dynamic and objective method for evaluating muscle function under constant angular velocity, enabling the quantification of parameters such as peak strength, total work, and muscular endurance.
Jump test for power | Baseline, 6 weeks, 12 weeks, and 8 weeks after detraining (up to 20 weeks per participant)
  Jump test by force platforms can provide multi-dimensional key parameters such as strength, power, speed and time by accurately measuring the ground reaction force (GRF).
Dance performance for the qualitative aspects | Baseline, 6 weeks, 12 weeks, and 8 weeks after detraining (up to 20 weeks per participant)
  The dance performance assessment was divided into two parts. The first part evaluated dance performance using the Performance Competence Evaluation Scale (PCEM); the intra- and inter-rater reliability coefficients were 0.95 and 0.94, respectively, indicating strong validity and reliability of the measure. The second part assessed competition performance based on the World Dancesport Federation (WDSF) rules, which are widely used in major dancesport competitions worldwide.

CONTACTS AND LOCATIONS:
Locations (1):
- Hubei normal university, Hubei, Huangshi, China

IPD SHARING:
Plan to Share IPD: Undecided